CLINICAL TRIAL: NCT00846144
Title: This Study is a Small Preliminary Study to Evaluate the Possibility of Performing a Phase 1 Study.
Brief Title: The Reduction in Glucose Stimulated Insulin Secretion Induced by Cytokines May be Prevented by Copper Addition - Studies in Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Prof. Itamar Raz, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0136-08-HMO
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Hyperglycemia; Diabetes
Keywords: Glucose stimulated insulin secretion; copper; cytokines; diabetes; Reduction in insulin secretion
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus | interventions — Copper Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: copper sulfate — copper sulfate 3mg/d for a period of 6 months

SUMMARY:
In the CDs rat model, beta-cell dysfunction and pancreatic exocrine damage are triggered and prevented by altering dietary Cu content suggesting a chronic and acute role for Cu. These abnormalities become apparent when the CDs rats are exposed to high sucrose low copper diet, triggering a vicious sequence of events: exocrine damage, recruitment of macrophages expressing IL-1beta leading to oxidative stress and even more reduction in the activity of Cu-dependent enzymes (chronic effect). When Cu levels are re-established (acute effect) they may prevent the inhibitory effect of IL-1beta on insulin release and may restore the activity of enzymes inhibited by IL-1beta. In this study we will identify humans with marginal Cu status that may benefit from copper supplementation to normalize their GSIS. These patients will be given a daily Cu supplement (3mg/d), or placebo for a period of 6 months. GSIS, pancreatic dysfunction and biomarkers of marginal Cu status will be measured in different blood components before and every 4 weeks during treatments or placebo.

ELIGIBILITY:
Inclusion Criteria:

* diabetic subjects with BMI < 33
* HbA1C < 8
* plasma copper levels of < 90 ul/dl

Exclusion Criteria:

* patients with bad physical conditions

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-09 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Identify humans with marginal Cu status that may benefit from copper supplementation and normalize their GSIS. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Itamar Raz, Prof, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Diabetes Unit, Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Weksler-Zangen S, Raz I, Lenzen S, Jorns A, Ehrenfeld S, Amir G, Oprescu A, Yagil Y, Yagil C, Zangen DH, Kaiser N. Impaired glucose-stimulated insulin secretion is coupled with exocrine pancreatic lesions in the Cohen diabetic rat. Diabetes. 2008 Feb;57(2):279-87. doi: 10.2337/db07-0520. Epub 2007 Oct 31. PMID 17977959
- [Background] Weksler-Zangen S, Yagil C, Zangen DH, Ornoy A, Jacob HJ, Yagil Y. The newly inbred cohen diabetic rat: a nonobese normolipidemic genetic model of diet-induced type 2 diabetes expressing sex differences. Diabetes. 2001 Nov;50(11):2521-9. doi: 10.2337/diabetes.50.11.2521. PMID 11679430